CLINICAL TRIAL: NCT03683589
Title: Contribution of De Novo Lipogenesis in Severity of Nonalcoholic Fatty Liver Disease
Brief Title: De Novo Lipogenesis in Severity of NAFLD
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Society for Nutrition (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, University of Missouri-Columbia
Other Study IDs: 2012544; R01DK113701 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2020-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Bariatric Surgery Candidate; Obesity, Morbid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be stored in a -80C freezer. Liver samples will be tested immediately and will not be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Participants will receive deuterated water for 10 days before undergoing bariatric surgery.
  Liver biopsy collected, lipids extracted and DNL measured via GC/MS.

SUMMARY:
NAFLD is the most prevalent liver disease in the U.S., and there is a serious need to understand its progression to the advanced state, nonalcoholic steatohepatitis (NASH). Previous studies has shown that elevated de novo lipogenesis (DNL) is the unique, early event distinguishing patients with NAFLD from equally-obese subjects with low IHTG. The purpose of this study is to directly by measure DNL in human liver tissue and comparing it to liver histological scores from patient biopsies.

DETAILED DESCRIPTION:
The development of nonalcoholic fatty liver disease (NAFLD) progresses from a state of elevated intrahepatic triglycerides (IHTG) to liver inflammation, and ultimately, hepatic apoptosis and fibrosis. NAFLD is the most prevalent liver disease in the U.S., and there is a serious need to understand its progression to the advanced state, nonalcoholic steatohepatitis (NASH). Elevated de novo lipogenesis (DNL) is the unique, early event distinguishing patients with NAFLD from equally-obese participants with low IHTG. DNL is the process of liver synthesis of fatty acids (FAs) from carbohydrate. In humans, studies have shown that DNL significantly predicts the magnitude of IHTG, however, it is unknown whether the pathway plays a role in disease progression. Evidence supporting this concept includes the fact that the primary product of DNL is the saturated FA, palmitate, which in cell culture has been shown to significantly contribute to oxidative stress and inflammation. Recent rodent data show that upregulation of DNL through dietary supplementation of sucrose exacerbated the hepatotoxic effects of excess dietary FAs. A preliminary abstract presented by others at the 2017 Liver Meeting suggested that DNL may not be different between patients with low and high liver fibrosis, although these data were collected using an indirect measure of liver disease. Here, in the present study, the hypothesis will be tested directly by measuring DNL in human liver tissue and comparing it to liver histological scores (NAFLD Activity Score, NAS) from patient samples.

ELIGIBILITY:
Inclusion and exclusion criteria are similar to the criteria set by a larger project (NCT03151798).

Inclusion criteria:

* Men and women (pre and post-menopausal)
* Overweight/obese with BMI ≥ 25.9 or ≤ 50.0 kg/m2
* Characteristics of the metabolic syndrome, pre-diabetes (fasting glucose 100-125 mg/dL or 2h glucose 140-200 mg/dL) or diabetes type II
* 22-65 years of age
* use of tobacco products or no use of these products
* Sedentary, ≤ 60 minutes per week of structured physical activity

Exclusion criteria:

• The following conditions exclude subjects for this project because bariatric surgery would not be performed in these populations. Individuals with acute disease or advanced cardiac, liver, or renal disease, excessive alcohol use, anticoagulation therapy, or any severe co-morbid condition limiting life expectancy < 1 year. Women pregnant or trying to become pregnant.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes both obese men and women who are undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
De novo lipogenesis | Dec 2019
  DNL will be measured directly in the liver biopsies

SECONDARY OUTCOMES:
Histological scores (NAFLD activity score) | Dec 2019
  Tissue histology will be performed to obtain NAFLD activity score (NAS). A pathologist, trained in determining the NAS of histological samples, grades them for the quantity of fat present, and the levels of inflammation and fibrosis. A score of 0 is considered completely healthy (devoid of any of these three characteristics), while a score of 8 indicates severe pathology, advanced as far as cirrhosis.
Liver enzymes | Dec 2019
  AST and ALT will be measured on the day when liver biopsy is collected
FibroScan | Dec 2019
  Liver fat and fibrosis will also be measured non-invasively via FibroScan TM

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lambert JE, Ramos-Roman MA, Browning JD, Parks EJ. Increased de novo lipogenesis is a distinct characteristic of individuals with nonalcoholic fatty liver disease. Gastroenterology. 2014 Mar;146(3):726-35. doi: 10.1053/j.gastro.2013.11.049. Epub 2013 Dec 4. PMID 24316260
- [Background] Donnelly KL, Smith CI, Schwarzenberg SJ, Jessurun J, Boldt MD, Parks EJ. Sources of fatty acids stored in liver and secreted via lipoproteins in patients with nonalcoholic fatty liver disease. J Clin Invest. 2005 May;115(5):1343-51. doi: 10.1172/JCI23621. PMID 15864352
- [Derived] Syed-Abdul MM, Moore MP, Wheeler AA, Ganga RR, Diaz-Arias A, Petroski GF, Rector RS, Ibdah JA, Parks EJ. Isotope Labeling and Biochemical Assessment of Liver-Triacylglycerol in Patients with Different Levels of Histologically-Graded Liver Disease. J Nutr. 2023 Dec;153(12):3418-3429. doi: 10.1016/j.tjnut.2023.09.018. Epub 2023 Sep 27. PMID 37774841